CLINICAL TRIAL: NCT04001426
Title: Pilot Phase for an Acute Evaluation of a Non-Implantable Electrical Continence Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FemPulse Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-003
Record Dates: First submitted 2019-06-24; First posted 2019-06-28 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive Bladder; Women; Neuromodulation; Bioelectronic Medicine
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Subjects will wear a device and will be monitored non-invasively during activation of the device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Monitoring during activation of the FemPulse System (Experimental): Subjects will undergo non-invasive monitoring during activation of the FemPulse System.
  Interventions: Device: The FemPulse System

INTERVENTIONS:
Device: The FemPulse System — Non-invasive monitoring during activation of the FemPulse System

SUMMARY:
The purpose of this feasibility clinical investigation is to investigate a new medical device treatment for Overactive Bladder (OAB) in women.

DETAILED DESCRIPTION:
The FemPulse System is a vaginal ring intended to provide mild electrical stimulation to nerves that regulate bladder function. It is believed that stimulation of these nerves may help relieve the symptoms of OAB.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy women ≥ 21 years old
* Using contraception if of reproductive age

Exclusion Criteria:

* Pregnant, recently pregnant or actively trying to conceive
* Prior hysterectomy
* Current or recent urinary tract or vaginal infection

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Autonomic nervous system response | Up to 6 hours
  The Quantitative Sudomotor Axon Reflex Test (QSART) will be used to detect changes in autonomic nervous system activity during device activation
Evoked Potential response | Up to 6 hours
  Surface electrodes will be used to detect whether evoked potentials are generated during device activation

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin Healthcare, Minneapolis, Minnesota, United States